CLINICAL TRIAL: NCT00361881
Title: A Randomized, Double-Blind, Active Controlled, Vehicle-Controlled, Subject Initiated Study Comparing Efficacy and Safety of ME-609 Versus Acyclovir Cream for Treatment of Recurrent Herpes Simplex Labialis
Brief Title: Efficacy and Safety Study of ME-609 and Acyclovir for Treatment of Herpes Simplex Labialis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medivir (Industry)
Responsible Party: Börje Darpö, MD, PhD, Medivir AB
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 609-04
Record Dates: First submitted 2006-08-08; First posted 2006-08-09 (Estimated); Last update posted 2008-08-18 (Estimated); Status verified 2008-08

CONDITIONS: Herpes Labialis
MeSH Terms: conditions — Herpes Labialis | interventions — ME 609; Acyclovir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): ME-609
  Interventions: Drug: ME-609
- 2 (Active Comparator): Acyclovir in ME-609 vehicle
  Interventions: Drug: acyclovir in ME-609 vehicle
- 3 (Placebo Comparator): Vehicle
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: ME-609 — Cream, dose 5 times daily during 5 days.
  Arms: 1
Drug: acyclovir in ME-609 vehicle — Dose 5 times daily for 5 days
  Arms: 2
Drug: Vehicle — Dose 5 times daily for 5 days
  Arms: 3

SUMMARY:
The purpose of this study is to determine whether ME-609 is more efficient than acyclovir and placebo for the treatment of recurrent herpes labialis.

DETAILED DESCRIPTION:
This was a randomized, double-blind, active- and vehicle-controlled study comparing the effects of ME-609, acyclovir in ME-609 vehicle, and vehicle alone. Treatment was subject-initiated within 1 hour of experiencing the first signs or symptoms of a herpes recurrence. The subject visited a study clinic as soon as possible after treatment initiation, but no later than midnight of the following day, for evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Generally good health
* History of recurrent herpes labialis with at last three episodes during the prior 12 months

Exclusion Criteria:

* Treatment with antivirals or immunosuppressive agents within 2 weeks prior to randomization
* Pregnant and/or nursing women
* Continuous daily treatment with pain medication
* Significant skin condition that occur in the area of herpes recurrences

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1443 (Actual)
Dates: Start 2006-07; Primary Completion 2007-08 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with non-ulcerative recurrences measured as the proportion of subjects in whom the study recurrence did not progress beyond the papule stage. | 5 days

SECONDARY OUTCOMES:
Episode duration | until healing

CONTACTS AND LOCATIONS:
Overall Officials: Christopher M Hull, MD, Principal Investigator
Locations (1):
- Coastal Caroline Research Center, Mt. Pleasant, South Carolina, United States

REFERENCES:
- [Derived] Hull CM, Harmenberg J, Arlander E, Aoki F, Bring J, Darpo B, Levin MJ, Tyring S, Spruance SL; ME-609 Study Group. Early treatment of cold sores with topical ME-609 decreases the frequency of ulcerative lesions: a randomized, double-blind, placebo-controlled, patient-initiated clinical trial. J Am Acad Dermatol. 2011 Apr;64(4):696.e1-11. doi: 10.1016/j.jaad.2010.08.012. Epub 2010 Sep 20. PMID 20851499